CLINICAL TRIAL: NCT05811039
Title: Efficacy and Safety of Remo-Wax® Oil (RWO) in Subjects With Isolated Itching of the External Ear Canal; an Open, Single-arm, Non-randomised, Multicentre Clinical Study
Brief Title: Efficacy and Safety of Remo-Wax® Oil (RWO) in Subjects With Isolated Itching of the External Ear Canal
Acronym: Remo_Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3126002
Record Dates: First submitted 2023-03-14; First posted 2023-04-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-05

CONDITIONS: Itching
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: Open, single-arm, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment with RemoWax Oil
  Interventions: Device: Remo-Wax® Oil

INTERVENTIONS:
Device: Remo-Wax® Oil — Remo-Wax® Oil (abbreviated RWO; GMDN (Global Medical Device Nomenclature) code 46259, Earwax softening oil), is a CE-marked, non-sterile fluid mixture, used for prevention of impacted earwax. Remo-Wax® Oil also moisturizes the skin in the ear canal and reduces itching and irritation caused by the ear canal dryness

SUMMARY:
Open, single-arm, non-randomized study to demonstrate the efficacy of Remo-Wax® Oil (abbreviated RWO) in the treatment of isolated itching of the external ear canal and to demonstrate the safety of the product.

DETAILED DESCRIPTION:
The study includes a 4-week treatment period with RWO. The first administrations are performed at the study site (Screening/Day 1). Thereafter, the doses are self-administered by the subjects once a day for 2 weeks (Days 2-14) and subsequently, RWO is self-administered once a week for two weeks, i.e. on Days 21 and 28. The subjects may take additional doses as needed at any time point during the treatment period. Final assessments will be performed at the End-of-Study Visit 1-3 days after the last RWO administration.

Itching of the ear canals will be assessed with questionnaires at the Screening and End-of-Study Visits. Irritation will be assessed by the ENT (ear-nose-throat) examination at the Screening and End-of-Study Visits. Satisfaction with the treatment procedure will be assessed with a questionnaire at the End-of-Study Visit. The subjects are keeping a study diary to document RWO administrations (as scheduled and potential additional doses), potential deviations from study-related instructions, AEs and device deficiencies (DD).

ENT examination including otomicroscopy will be performed at Screening and End-of-Study Visits. AEs and DDs will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent obtained.
2. ≥12 years old male or female subjects who, in the opinion of the Investigator, are able to comply with the study procedures and evaluations
3. Subjects with complaints of recurrent or continuous unilateral or bilateral itchy ear canals
4. A score of at least 5 in subjective pruritus evaluation using a score of itching between 0 (none) and 10 (extreme) in the ear canal at its worst in the previous four days
5. No ear-related abnormal findings in an ENT examination by an otolaryngologist, with the exception that mild to moderate irritation in the ear canal is allowed
6. For participants who are minors: A representative/caregiver (per local requirements) available, who provides the Informed Consent on behalf of the minor subject and who is accompanying the subject at the study visits, as relevant, and supports the subject with home administrations and filling in the study diary, as relevant

Exclusion Criteria:

1. Hypersensitivity to any product ingredient(s) or history of anaphylactic/anaphylactoid reactions
2. History of tympanic membrane perforation or tympanostomy tubes in the previous 6 months
3. External ear or ear canal infection/inflammation in the previous 30 days
4. Otitis media/myringitis in the previous 30 days
5. Past ear surgery
6. Otorrhea in the previous 30 days
7. Temporal bone neoplasm
8. Presence of known or suspected mastoiditis
9. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data (e.g. impacted cerumen, ear eczema or seborrhoea, ear canal stenosis, exostoses).
10. Subjects with a history of long-term topical or systemic steroid and/or antibiotic use (according to Investigator's judgement), and those who had used topical or systemic steroids and/or antibiotics in the previous 30 days
11. Subjects with systemic disease such as diabetes mellitus, renal or hepatic disorders, or dermatological disease such as psoriasis or atopic dermatitis
12. Participation in a clinical drug study or another clinical investigation within 60 days prior to the start of the present study
13. Subjects who are not able to perform the administrations by themselves

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Itchiness | The itching score is filled in by the subject at Screening Visit and at the End-of-Study Visit (conducted 4 weeks later). As an average, a decline of at least 2.5 scores is required for the RWO to be considered efficacious.
  Primary efficacy evaluation is based on subjective pruritus evaluation using a Visual Analogue Scale (VAS) score of itching in the ear canal between 0 (none) and 10 (extreme).

SECONDARY OUTCOMES:
Irritation | From Screening to End-of-Study Visit (4 weeks later).
  Only those subjects with irritation at screening will be evaluated for this endpoint. For this analysis, the ears will be evaluated separately (not by subject) in the Ear-Nose-Throat (ENT) examination. The assessment will grade the irritation in the ear canal(s) as mild/moderate/severe and the analysis will look at the change in grade between the two assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Vilnius University Hospital, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No